CLINICAL TRIAL: NCT06420440
Title: Efficacy and Safety of Neoadjuvant HAIC Combined With Tislelizumab and Lenvatinib in Patients With Resectable HCC Screened by a Multimodal Deep Learning Model: a Multicenter Randomized Controlled Trial.
Brief Title: Neoadjuvant Therapy in Patients With Resectable HCC Screened by a Multimodal Deep Learning Model
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chen Xiaoping (Other)
Responsible Party: Sponsor-Investigator, Chen Xiaoping, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Neoadj-Net01
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: HCC
Keywords: Hepatocellular carcinoma; Neoadjuvant tehrapy; recurrence; Deep learning
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence | interventions — lenvatinib; tislelizumab; Hepatectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant therapy group (Experimental): Patients in the neoadjuvant group received neoadjuvant therapy prior to surgery (two cycles of HAIC combined with Tislelizumab and Lenvatinib), and adjuvant therapy (Tislelizumab for 8 cycles) after surgery.
  Interventions: Procedure: Hepatic arterial infusion chemotherapy; Drug: Lenvatinib; Drug: Tislelizumab; Procedure: Liver resection
- Direct liver resection group (Active Comparator): Patients in the control group underwent liver resection directly and received adjuvant therapy (Tislelizumab for 8 cycles) after surgery.
  Interventions: Procedure: Liver resection; Drug: Tislelizumab

INTERVENTIONS:
Procedure: Hepatic arterial infusion chemotherapy — Patients in the neoadjuvant group received two cycles of neoadjuvant hepatic arterial infusion chemotherapy (HAIC, adoption of the FOFOLX6 program, Folinic acid+5-fluorouracil+Oxaliplatin, 21 days between second HAIC treatments with a window of ±3 days)
  Arms: Neoadjuvant therapy group
Drug: Lenvatinib — Patients in the neoadjuvant therapy group received Lenvatinib before surgery(Len was started before HAIC treatment, discontinued during HAIC treatment, and discontinued approximately two weeks before surgery, Oral 8 mg or 12mg once a day depending body weight).
  Arms: Neoadjuvant therapy group
Drug: Tislelizumab — Patients in the neoadjuvant therapy group received two cycles of Tislelizumab therapy before surgery (First treatment with Tislelizumab was started 0-1 days after HAIC, 200 mg IV, followed by a second treatment 21 days later)
  Arms: Neoadjuvant therapy group
Procedure: Liver resection — Patients in the neoadjuvant therapy group were evaluated for tumor status and surgical safety after neoadjuvant therapy, and eligible patients subsequently underwent surgical resection. Patients in the direct surgery group underwent liver resection.
Drug: Tislelizumab — Given the high risk of postoperative recurrence, patients in both groups received adjuvant Tis therapy (every 21 days for 8 cycles) starting about one month after surgery.

SUMMARY:
Primary liver cancer is one of the most common malignant tumors in the world, and about 80%~90% of primary liver cancers are pathologically characterized as hepatocellular carcinoma (HCC). Radical surgery is the main method for patients with HCC to obtain long-term survival. However, the early recurrence rate of high-risk HCC is very high, which seriously affects the overall therapeutic effect.

DETAILED DESCRIPTION:
The protocol was revised in April 2025 (V1.1). Primary liver cancer is one of the most common malignant tumors in the world, and about 80%~90% of primary liver cancers are pathologically characterized as hepatocellular carcinoma (HCC). Radical surgery is the main method for patients with HCC to obtain long-term survival. However, the early recurrence rate of high-risk HCC is very high, which seriously affects the overall therapeutic effect. Although the tumor is in BCLC-A stage, when the tumor diameter is more than 5cm, the effect of surgery is worse than that of single small HCC due to the large resection range, the high risk of surgery and residual disease. In addition, BCLC-stage B and C tumors have a high recurrence rate due to multiple lesions or macrovascular invasion. To address this issue, new tools are urgently needed to guide the selection of appropriate treatment regimens to reduce the risk of postoperative recurrence and improve overall survival.

The investigators multidisciplinary team used deep learning technology to construct an artificial intelligence prediction model of neoadjuvant therapy (Neoadj-Net) benefit based on pre-treatment genetic testing data, digital pathology slides and imaging data (enhanced MRI) of 536 intermediate-stage HCC patients treated with HAIC in combination with lenvatinib and PD-1 monoclonal antibody in six centers, and external center data validated the model's good ability to identify the beneficiary population of the combination regimen ( AUC 0.89, Accuracy 0.86). This study is to explore the effectiveness and safety of Neoadj-Net in reducing postoperative recurrence by observing the benefit of the combined neoadjuvant regimen in patients who are potentially benefited from neoadjuvant therapy and direct surgery from the perspective of precision therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75.
2. No previous local or systemic treatment for hepatocellular carcinoma.
3. Child-Pugh liver function score ≤ 7.
4. ECOG PS 0-1.
5. No serious organic diseases of the heart, lungs, brain, kidneys, etc.
6. Enhanced MRI determines that the tumor is technically resectable but at high risk for recurrence(BCLC-A tumor diameter more than or equal to 5cm; BCLC-B; BCLC-C) ; without distant metastasis.
7. Pathologic type of hepatocellular carcinoma confirmed by puncture biopsy.
8. Multimodal Deep Learning Model Screening Based on Pathology, Imaging, and Genetic Data Suggests Benefit from HAIC in Combination with Lenvatinib and PD-1 inhibitors.

Exclusion Criteria:

1. Pregnant and lactating women.
2. Suffering from a condition that interferes with the absorption, distribution, metabolism, or clearance of the study drug (e.g., severe vomiting, chronic diarrhea, intestinal obstruction, impaired absorption, etc.).
3. A history of gastrointestinal bleeding within the previous 4 weeks or a definite predisposition to gastrointestinal bleeding (e.g., known locally active ulcer lesions, fecal occult blood ++ or more, or gastroscopy if persistent fecal occult blood +) that has not been targeted, or other conditions that may have caused gastrointestinal bleeding (e.g., severe fundoplication/esophageal varices), as determined by the investigator.
4. Active infection.
5. Other significant clinical and laboratory abnormalities that affect the safety evaluation.
6. Inability to follow the study protocol for treatment or follow up as scheduled.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Median event-free survival (EFS) | From date of randomization until the date of first documented recurrence or date of death from any cause, whichever came first, assessed up to 60 months.
  EFS is defined as the time from randomization to disease recurrence and/or disease progression or death from any cause.

SECONDARY OUTCOMES:
Safety Assessment | Baseline up to 12 months
  Any adverse event during treatment that is incompatible with the therapeutic purpose of the medication.The incidence and severity of adverse events and serious adverse events as assessed by CTCAE v5.0.
Overall Survival (OS) | From date of randomization until the date of death from any cause, assessed up to 60 months.
  OS is defined as the time from randomization to death from any cause

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Huapeng Sun, Xiangyang, Hubei
  - Enyu Liu, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: No